CLINICAL TRIAL: NCT07169500
Title: Clinical Study on the Safety and Efficacy of Autologous Hematopoietic Stem Cell Transplantation Combined With BCMA-CART in the Treatment of Young and Newly Diagnosed Multiple Myeloma
Brief Title: Autologous Transplantation Combined With BCMA CAR-T in the Treatment of Young NDMM
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Hebei Taihe Chunyu Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025025
Record Dates: First submitted 2025-07-31; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BCMA CART (Experimental): The subject underwent ASCT and BCMA-CART infusion
  Interventions: Biological: CAR-T

INTERVENTIONS:
Biological: CAR-T — Chimeric antigen receptor T cells (car-t) are genetically engineered MHC independent tumor specific killer cells.

SUMMARY:
To evaluate the safety and efficacy of autologous hematopoietic stem cell transplantation (ASCT) combined with BCMA-CART in the treatment of young NDMM

DETAILED DESCRIPTION:
This study is a single center, prospective clinical study initiated by researchers to evaluate the safety and efficacy of autologous hematopoietic stem cell transplantation combined with BCMA-CART cells in the treatment of young patients with newly diagnosed multiple myeloma, aiming to explore the safety and efficacy of ASCT combined with BCMA-CART in the treatment of young patients with NDMM.

ELIGIBILITY:
Inclusion Criteria:

Young newly diagnosed multiple myeloma (NDMM), 18-50 years old, suitable for ASCT;

1. The subjects voluntarily participated in the study and signed the informed consent form (ICF) by themselves or their legal guardians;
2. The subject must have proper organ function and meet all the following inspection results:

   total serum bilirubin (TBIL) ≤ 1.5 times the upper limit of normal (ULN); serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN; creatinine clearance (CrCl) (Cockcroft Gault formula) ≥ 40ml/min; prothrombin time (PT) ≤ 1.5 × ULN, partial prothrombin time (APTT) < 1.5 × ULN; international normalized ratio (INR) < 1.5 × ULN; hemoglobin (HB) ≥ 60g/L; absolute neutrophil count (ANC) ≥ 1.0 × 10^9/lL(no growth factors such as granulocyte colony stimulating factor [G-CSF] have been received within 7 days before the laboratory examination in the screening period); absolute lymphocyte count (ALC) ≥ 0.5 × 10^9/L; platelet (PLT) ≥ 50 × 10^9/L (no platelet transfusion within 7 days before the laboratory examination in the screening period); left ventricular ejection fraction (LVEF) ≥ 45%; blood oxygen saturation (SpO2) ≥ 92%;
3. The ECOG score is 0-1. See Appendix V for ECOG score;
4. Estimated survival ≥ 3 months;
5. The pregnancy test of fertile female subjects should be negative and not during lactation.

Exclusion Criteria:

1. Have a history of allergy to any component in cell products;
2. Serious heart disease, including but not limited to:

   myocardial infarction, cardiac angioplasty or stent implantation within 6 months before signing ICF; unstable angina; severe arrhythmia; history of severe non ischemic cardiomyopathy; congestive heart failure (New York Heart Association [NYHA] class III or IV), see Appendix II for NYHA score;
3. History of autologous / allogeneic hematopoietic stem cell transplantation;
4. Stroke or seizure within 6 months before signing ICF;
5. Have autoimmune diseases, immunodeficiency or other diseases that need immunosuppressant treatment;
6. Within 3 years before signing the ICF, patients with malignant tumors other than multiple myeloma, except for fully treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, local prostate cancer after radical surgery, breast ductal carcinoma in situ after radical surgery, and carcinoma in situ in other parts one year after radical surgery, and there has been no treatment and no sign of recurrence in the screening period;
7. The presence of uncontrolled active infection;
8. Unstable systemic diseases judged by the investigator: including but not limited to serious liver, kidney or metabolic diseases requiring drug treatment;
9. One week before lymphocyte collection, the memory is under any of the following conditions:

the detection value of hepatitis B virus (HBV) DNA in peripheral blood is higher than the lower limit of detection; hepatitis C virus (HCV) antibody positive and peripheral HCV-RNA positive.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2028-03-02 (Estimated); Study Completion 2030-03-02 (Estimated)

PRIMARY OUTCOMES:
MRD negative rate at 3 month after the treatment of autologous transplantation combined with CART. | 3 month
  MRD by flow cytometry

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | 2 years after CAR-T infusion
  Time from CAR-T infusion to first documentation of progressive disease (PD), or death due to any cause, whichever occurs first
Minimal Residual Disease (MRD) negetive rate | at day28, M2, M3, M6, M9, M12, M15, M18, M24 after CAR-T infusion
  Proportion of subjects who achieved MRD negative
Overall response rate (ORR) evaluated by the investigators | 2 years after CAR-T infusion
  Percentage of subjects who achieved partial response (PR) or better according to IMWG Uniform Response Criteria for Multiple Myeloma as assessed by the investigators
Duration of Response (DOR) | 2 years after CAR-T infusion
  Time from first response evaluated by an investigators to disease progression or death from any cause
Time to Response (TTR) | 2 years after CAR-T infusion
  Time from CAR-T infusion to first documentation of response evaluated by an investigator
Overall Survival (OS) | 2 years after CAR-T infusion
  Time from CAR-T infusion to time of death due to any cause
PK:Cmax,Tmax,AUC(0-28days),Tlast | 2 years
  flow cytometry and qPCR

CONTACTS AND LOCATIONS:
Overall Officials: Yan Xu, MD, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No